CLINICAL TRIAL: NCT03432455
Title: Incidence and Prevalence of Juvenile Dermatomyositis in Alsace Between 2000 to 2015
Brief Title: Incidence and Prevalence of Juvenile Dermatomyositis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6784
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Juvenile Dermatomyositis
Keywords: Incidence; prevalence; epidemiology; juvenile dermatomyositis; inflammatory myopathy
MeSH Terms: conditions — Dermatomyositis; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive, retrospective, multi-center, cross-sectional and observational epidemiological study of incidence and prevalence of juvenile dermatomyositis in Alsace from 2000 to 2015. Alsace is a French region with a low migratory flow

ELIGIBILITY:
Inclusion Criteria:

* Age under 16 years
* Have a dermatomyositis according to the diagnostic criteria of Bohan and Peter of 1975

Exclusion Criteria:

* Refusal to participate in the study

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: Patient who have a dermatomyositis according to the diagnostic criteria of Bohan and Peter of 1975
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Identify incident and prevalent cases of juvenile dermatomyositis according to Bohan and Peter's criteria at january 1st, 2016 via capture/recapture strategy | The period from from January 1st, 2000 to December 31st, 2015 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, Strasbourg, France